CLINICAL TRIAL: NCT06902207
Title: Real-life Incidence of Intraocular Inflammation Following Intravitreal Faricimab Therapy
Brief Title: Real-world Incidence of Intraocular Inflammation Following Intravitreal Faricimab Therapy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: p-2024-16902
Record Dates: First submitted 2025-03-15; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Intraocular Inflammation
Keywords: faricimab; intravitreal injection; anti-VEGF; intraocular inflammation
MeSH Terms: conditions — Uveitis | interventions — faricimab; Intravitreal Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Faricimab Injection [Vabysmo] — The procedures followed local standard protocol, that included the use of 2-3 drops of topical tetracaine anesthesia, use of an eye speculum, topical 5% povidone-iodine disinfection, 33G-needle, injection site 3.5 mm posterior from the limbus marked by calipers in the supertemporal or the inferotemporal quadrant, sterile cotton tip tamponade at the site of injection after removal of the needle, and no post-procedure antibiotics.
  Other Names: Intravitreal injection

SUMMARY:
Faricimab (Vabysmo®), a novel pharmaceutical agent is a promising treatment for age-related macular degeneration and diabetic macular edema due to its dual mechanism of action, targeting both the VEGF and angiopoietin-2 (Ang-2) pathways, offering potential benefits in improving visual outcomes and reducing treatment burdens. The phase 3 TENAYA and LUCERNE clinical trials have demonstrated its efficacy and safety profile, leading to regulatory approval and increasing use in clinical practice. However, as with any new therapeutic agent, there is a critical need to monitor and evaluate real-world safety data to complement and validate clinical trial findings.

Intraocular inflammation (IOI), which is a significant adverse effect of intravitreal anti-VEGF injections, is of particular interest as it can vary from a mild transient reaction to a potentially vision-threatening outcome.

The incidence and severity of IOI in a real-world settings can vary from clinical trial results due to differences in patient populations, injection techniques, and clinical settings.

The aim of this study is to estimate the real-life incidence of intraocular inflammation following intravitreal faricimab injections at a large, regional highly specialized tertiary center.

ELIGIBILITY:
Inclusion criteria

* >18 years of age
* Having received at least 1 intravitreal faricimab injection at our center
* Follow-up period of at least 6 weeks after the injection

Exclusion criteria for IOI cases

* Having received intravitreal injections of other types (e.g., intravitreal steroids, antiviral agents) at the same time as the intravitreal anti-VEGF injection or during the follow-up period
* Underwent intraocular surgery within 6 weeks before or after the intravitreal injection, except for surgical interventions that are meant to diagnose or treat the actual IOI in question (e.g., diagnostic chamber tap, diagnostic vitrectomy, vitrectomy for suspected endophthalmitis, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Capital Region of Denmark who are receiving faricimab injections at our center.
Sampling Method: Non-Probability Sample
Enrollment: 6053 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of intraocular inflammation (IOI) | 01/NOV/2023 - 31/AUG/2024
  Incidence of IOI following the faricimab injection procedure, described as cases per eye, cases per patient and cases per injection

SECONDARY OUTCOMES:
Differences in age | 01/NOV/2023 - 31/AUG/2024
  Between individuals developing and not developing IOI following faricimab injection
Differences in sex | 01/NOV/2023 - 31/AUG/2024
  Between individuals developing and not developing IOI following faricimab injection
Differences in number of anti-VEGF injections | 01/NOV/2023 - 31/AUG/2024
  Between individuals developing and not developing IOI following faricimab injection
Differences between treatment-naïve and switch-patients | 01/NOV/2023 - 31/AUG/2024
  Differences in developing and not developing IOI following faricimab injection between patients that received previous anti-VEGF treatments before faricimab and those that did not.
Time from injection to onset of IOI | 01/NOV/2023 - 31/AUG/2024
  Measured in days
Disease duration of IOI | 01/NOV/2023 - 31/AUG/2024
  Measured in days
Functional outcome of IOI cases | 01/NOV/2023 - 31/AUG/2024
  Best-corrected visual acuity (BCVA) before, at, and after onset of the IOI. Measured in Snellen acuity, converted to logMAR.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Rigshospitalet, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] Anderson WJ, da Cruz NFS, Lima LH, Emerson GG, Rodrigues EB, Melo GB. Mechanisms of sterile inflammation after intravitreal injection of antiangiogenic drugs: a narrative review. Int J Retina Vitreous. 2021 May 7;7(1):37. doi: 10.1186/s40942-021-00307-7. PMID 33962696
- [Background] Fine HF, Despotidis GD, Prenner JL. Ocular inflammation associated with antivascular endothelial growth factor treatment. Curr Opin Ophthalmol. 2015 May;26(3):184-7. doi: 10.1097/ICU.0000000000000154. PMID 25822254
- [Background] Shirley M. Faricimab: First Approval. Drugs. 2022 May;82(7):825-830. doi: 10.1007/s40265-022-01713-3. PMID 35474059
- [Background] European Medicines Agency (2022) Vabysmo. https://www.ema.europa.eu/en/medicines/human/EPAR/vabysmo Accessed: 07 Sep 2023
- [Background] Heier JS, Khanani AM, Quezada Ruiz C, Basu K, Ferrone PJ, Brittain C, Figueroa MS, Lin H, Holz FG, Patel V, Lai TYY, Silverman D, Regillo C, Swaminathan B, Viola F, Cheung CMG, Wong TY; TENAYA and LUCERNE Investigators. Efficacy, durability, and safety of intravitreal faricimab up to every 16 weeks for neovascular age-related macular degeneration (TENAYA and LUCERNE): two randomised, double-masked, phase 3, non-inferiority trials. Lancet. 2022 Feb 19;399(10326):729-740. doi: 10.1016/S0140-6736(22)00010-1. Epub 2022 Jan 24. PMID 35085502
- [Background] Khanani AM, Patel SS, Ferrone PJ, Osborne A, Sahni J, Grzeschik S, Basu K, Ehrlich JS, Haskova Z, Dugel PU. Efficacy of Every Four Monthly and Quarterly Dosing of Faricimab vs Ranibizumab in Neovascular Age-Related Macular Degeneration: The STAIRWAY Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2020 Sep 1;138(9):964-972. doi: 10.1001/jamaophthalmol.2020.2699. PMID 32729897